CLINICAL TRIAL: NCT03679130
Title: FitMum: Fitness for Good Health of Mother and Child
Acronym: FitMum-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Technical University of Denmark (Other); University of Aarhus (Other); University of Graz (Other); Deakin University (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ellen Christine Leth Loekkegaard, Professor, Chief Physician, PhD, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-18011067
Record Dates: First submitted 2018-08-30; First posted 2018-09-20 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy Related; Physical Activity
Keywords: Pregnancy; Physical activity; Healthy; Epigenetics; Process evaluation; Doubly labeled water
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: FitMum RCT is designed as an open-labeled single-site three-arm randomized controlled trial, including 220 pregnant women no later than gestational age week 15+0 days. Included women will be randomized in a 2:2:1 ratio to receive a structured supervised exercise training (EXE) intervention, receive a motivational counseling intervention supported by health technology (MOT), or a control group receiving standard treatment (CON), respectively. The participants in the EXE and MOT groups continue in the physical activity intervention as long as their pregnancy allows and ideally until delivery, in total approximately six months. Collection of data for assessment of the primary outcome will take place from randomization (one week after inclusion) to GA week 28+0-6 and will be measured by a commercial activity tracker. Secondary outcomes will be examined at Nordsjaellands Hospital six times during the study period. Time frames and methods for assessment of outcomes are specified below.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured exercise training (EXE) (Experimental): Structured supervised exercise training (EXE) contains three weekly one-hour exercise sessions at moderate intensity, more specifically one water exercise session and two land exercise sessions. The training will be supervised, held in teams, and both water and land exercise sessions will consist of a combination of aerobic and resistance training.
  Interventions: Behavioral: Structured supervised exercise training
- Motivational counseling (MOT) (Experimental): Motivational counseling supported by health technology (MOT) contains four individual and three group counseling sessions taking place from randomization until GA week 33+6 and aim to motivate the participants to increase their physical activity level at moderate intensity. During individual sessions, feedback on physical activity performance will be provided based on activity data acquired from the activity tracker and further, MOT-participants will receive weekly SMS-reminders about physical activity.
  Interventions: Behavioral: Motivational counseling supported by health technology
- Control group (CON) (No Intervention): Control group receiving standard treatment.

INTERVENTIONS:
Behavioral: Structured supervised exercise training — EXE contains three weekly one-hour exercise sessions at moderate intensity, more specifically one water exercise session and two land exercise sessions. The training will be supervised, held in teams, and both water and land exercise sessions will consist of a combination of aerobic and resistance training.
  Other Names: EXE
  Arms: Structured exercise training (EXE)
Behavioral: Motivational counseling supported by health technology — MOT contains four individual and three group counseling sessions taking place from randomization until GA week 33+6 and aim to motivate the participants to increase their physical activity level at moderate intensity. During individual sessions, feedback on physical activity performance will be provided based on activity data acquired from the activity tracker and further, MOT-participants will receive weekly SMS-reminders about physical activity.
  Other Names: MOT
  Arms: Motivational counseling (MOT)

SUMMARY:
A physically active lifestyle during pregnancy has potential to improve maternal and child health. However, less than four out of ten Danish pregnant women succeed to achieve 30 minutes of daily physical activity at moderate intensity as recommended by the Danish Health Authorities. This project investigates how to implement physical activity in pregnant women´s everyday life by testing the efficacy of two very different exercise programs on physical activity level during pregnancy.

DETAILED DESCRIPTION:
Low levels of physical activity during pregnancy constitute a significant public health issue as increasing evidence suggests that the mother's lifestyle during pregnancy may influence the future health of her child. A physically active lifestyle during pregnancy has potential to improve metabolic health of mother and child and thus may play an important role in relation to counteracting the obesity epidemic and the increasing incidence of metabolic diseases that escalates globally.

However, less than four out of ten Danish pregnant women succeed to achieve 30 minutes of daily physical activity at moderate intensity as recommended by the Danish Health Authorities. The key gap in evidence and practice towards tackling the significant public health issue of being physically inactive during pregnancy is lack of evidence of how physical activity can be implemented. Only very few and scattered regional or municipal physical activity initiatives are currently targeting Danish pregnant women, and these are mainly targeted overweight women. Implementing and validating means to empower the pregnant women to be physically active have the potential to establish the norm of being physically active during pregnancy and might halt the negative spiral effect of physical inactivity, obesity and metabolic diseases that escalates globally.

The aim of FitMum RCT is to evaluate the effects of structured supervised exercise training and motivational counseling supported by health technology on physical activity level during pregnancy. The two exercise programs are designed to meet the motivators and overcome the specific barriers for physical activity among pregnant women. The programs will be tested in a three-armed randomized controlled trial including 220 healthy, physically inactive, pregnant women.

FitMum is carried out in collaboration between University of Copenhagen, Nordsjaellands Hospital, Technical University of Denmark, Aarhus University and international researchers.

During the COVID-19 pandemic supplies of interventions and test visits are periodically changed. During lockdown periods, all interventions and test visits (except delivery) are converted into online versions. In EXE, the water exercise sessions are replaced with online land exercises. All land exercise sessions consist of 30 min of aerobic exercise where the participants exercise on their own followed by 30 min of supervised online group resistance training. All individual and group MOT sessions are held online. As much data as possible is collected during the pandemic, but in some periods, biological samples and DXA scans have been cancelled and participants were weighed at home.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed
* Pregnant woman aged 18 years or older
* Gestational age of max. 15+0 weeks
* Ultrasonic confirmed intrauterine pregnancy
* BMI of 18.5-40 kg/m2 calculated from pre-pregnancy weight or first measured weight in pregnancy

Exclusion Criteria:

* Severe chronic disease
* Structured exercise at moderate to vigorous intensity more than 1 hour per week during pregnancy
* Previous preterm delivery (before GA week 37)
* Obstetric or medical complications
* Multiple pregnancies
* Non-Danish speaking
* Alcohol or drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — As only women can be pregnant, only women are eligible in participating in the interventional part of the study.
  However, we encourage the biological father of the child to consent on providing a paternal blood sample for epigenetic analysis.
Enrollment: 220 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Min/week of moderate-to-vigorous-intensity physical activity from randomization to GA week 28+0-6 determined by a Garmin Vivosport activity tracker [ Time Frame: Continuously 24/7 from inclusion (at latest GA week 15+0) to GA week 28+0-6 ]' | Continuously 24/7 from inclusion (at latest GA week 15+0) to GA week 28+0-6
  Physical activity level from randomization to GA week 28+0-6 determined by a wrist-worn activity tracker, Garmin Vivosport, with built-in heart rate monitor and accelerometer. The activity tracker is to be worn continuously by the women from inclusion until delivery. After inclusion baseline physical activity level will be measured for one week, followed by randomization to one of the three study groups and continuous monitoring of physical activity level by the activity tracker. Preferably, the activity tracker is also worn continuously from delivery and one year ahead. The activity tracker determines the frequency, duration and intensity of activity periods on a minute-to-minute basis and data from the activity tracker is wirelessly synced to its associated smartphone application, Garmin Connect, and research platform, Fitabase.

SECONDARY OUTCOMES:
Gestational weight gain | Baseline weight, weight at inclusion, weight at GA week 28+0-6, weight at GA 34+0-6 and weight at delivery.
  Weight gain during pregnancy
Complementary measures of physical activity level - by PPAQ-DK | At inclusion, GA week 28+0-6 and 34+0-6
  A Danish version of the validated 'Pregnancy Physical Activity Questionnaire' (PPAQ-DK) will be used to subjectively measure physical activity level during pregnancy.
Complementary measures of physical activity level - by doubly labeled water | At GA week 28+0-6
  The doubly labeled water technique will be used to measure free-living energy expenditure at GA week 28+0-6.
Complementary measures of physical activity level - by activity tracker | Continuously 24/7 from inclusion to delivery
  The activity tracker will also be used to measure physical activity level of the mother during the entire pregnancy period, meaning after GA week 28+0-6 until delivery as well.
Complementary measures of physical activity level - by activity tracker | Continuously 24/7 from delivery and one year ahead
  The activity tracker will also be used to measure physical activity level of the mother one year after delivery.
Clinical outcomes of mother and child | Delivery
  Clinical pregnancy, delivery and neonatal outcomes will be collected from medical records. E.g. incidence of Gestational Diabetes Mellitus, gestational age at delivery, mode of delivery, induction of labor, epidural, 5-minute Apgar score, pH of umbilical cord and birth weight.
Maternal body composition during pregnancy | At GA week 28+0-6
  Maternal body composition will be assessed by doubly labeled water during pregnancy.
Maternal body composition after delivery | One week after delivery
  Maternal body composition will be assessed by DXA scanning after delivery.
Maternal health-related quality of life and function | At inclusion, GA week 28+0-6, 34+0-6, and one year after delivery
  Health-related quality of life and function will be determined by a Danish version of the questionnaire "Medical Outcomes Study Short Form 36" (SF-36).
Maternal sick leave and pelvic and low back pain | At inclusion, GA week 28+0-6, and 34+0-6
  Sick leave and pelvic and low back pain will be assessed by a questionnaire verbally administered at interviews at visits.
Maternal sleep - by activity tracker | Continuously 24/7 from inclusion (at latest GA week 15+0) to 1 year after delivery
  Sleep quantity and quality will be assessed continuously by the activity tracker.
Maternal sleep - by PSQI | At inclusion, GA week 28+0-6, GA week 34+0-6 and one year after delivery
  Sleep quantity and quality will be assessed by a Danish version of the questionnaire "Pittsburgh Sleep Quality Index" (PSQI).
Metabolic markers in mother and child | At inclusion, GA week 28+0-6, 34+0-6, and delivery
  Plasma metabolites and hormones (e.g. triglyceride, HDL, LDL, total cholesterol and HbA1C) will be assessed by analysing maternal blood and umbilical cord blood.
DNA methylation | At GA week 34+0-6 and delivery.
  Epigenetic profiles will be assessed by analysing DNA methylation in maternal blood, paternal blood and umbilical cord blood.
Placental function | At delivery
  Placental function will be assessed via analyses of placental samples, maternal blood and umbilical cord blood.
Personal understandings of physical activity in everyday life - by qualitative interviews | From inclusion (at latest GA week 15+0) to delivery
  Investigations of personal understandings of physical activity in everyday life of pregnant women and social, structural and cultural practices and factors influencing successful implementation of exercise during pregnancy will be based on semi-structured qualitative interviews
Personal understandings of physical activity in everyday life - by observations | From inclusion (at latest GA week 15+0) to delivery
  Investigations of personal understandings of physical activity in everyday life of pregnant women and social, structural and cultural practices and factors influencing successful implementation of exercise during pregnancy. Data will be collected by observations
Personal understandings of physical activity in everyday life - by auto-documentation | From inclusion (at latest GA week 15+0) to delivery
  Investigations of personal understandings of physical activity in everyday life of pregnant women and social, structural and cultural practices and factors influencing successful implementation of exercise during pregnancy. Data will be collected by auto-documentation.
A process evaluation of FitMum RCT interventions | From inclusion (at latest GA week 15+0) to delivery
  Mixed methods will be used to do a qualitative and quantitative process evaluation. Data for the process evaluation are based on semi-structured qualitative interviews and administratively collected process data (e.g. frequency of training and counseling sessions, visits and measurements), electronic case report form files, and activity logs.
Physical activity behavior changes among pregnant women | At inclusion, GA week 28+0-6, GA week 34+0-6 and one year after delivery
  Self-efficacy for physical activity will be measured by a Danish version of the American questionnaire "Pregnancy Exercise Self-efficacy Scale" (P-ESES-DK).
Motivation for physical activity among pregnant women | At inclusion, GA week 28+0-6, GA week 34+0-6 and one year after delivery
  Motivation for physical activity will be measured by a Danish version of the British questionnaire "Behavioral Regulation Exercise Questionnaire" (BREQ-2).
Offspring growth in the first year of life | At 5 weeks, 5 months and 12 moths after delivery
  Growth in the offspring will be assessed by questionnaires, using data from visits to the participants' general practitioners.
Physical psycho-motor development in the offspring | One year after due date
  Physical psycho-motor development in the offspring will be assessed using a Danish version of the questionnaires Ages and Stages 3 (ASQ-3) for 12- and 14 month old babies.
Physical activity level in the offspring for 7 days, determined by a wrist band accelerometer Actigraph GT3X+ | One year after due date until one year and 7 days after due date
  Physical activity level one year after due date, determined by a wrist-worn accelerometer, Actigraph GT3X+. The activity tracker is to be worn continuously by offspring for 7 days. Data is stored in the device and transferred to the researchers' computer.
Mental well-being in mothers and fathers post partum | 6 weeks after delivery
  Mental well-being in mothers and fathers post partum will be assessed using a Danish validated screening-tool for parental post-partum depression, primarily based on the Edinburgh Postnatal Depression Scale and selected questions from The Masculine Depression Scale.
Validation of activity tracker, Garmin Vivosport, for measuring sleep | For one night, between GA week 28+0 until delivery
  validation of activity trackers for measuring sleep will be conducted using polysomnography (PSG) in a sub-group of forty women already participating in FitMum RCT. The women will wear the PGS for one night.
Breastmilk composition | 7-14 days after delivery
  Breastmilk for metabolomics and lipidomics analyses is obtained from one single feed 7-14 days after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Bente M Stallknecht, PhD, DMSc, Study Director — Department of Biomedical Sciences at University of Copenhagen; Ellen CL Løkkegaard, PhD, Principal Investigator — Department of Gynecology and Obstetrics at Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Undecided: It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Jessen AD, Alomairah SA, Jensen IKB, de Place Knudsen S, Roland CB, Bendix JM, Molsted S, Lokkegaard E, Stallknecht B. Mapping postpartum physical activity, sedentary time, and sleep: assessing the impact of prenatal physical activity interventions in the FitMum randomized controlled trial. Sci Rep. 2025 Oct 3;15(1):34606. doi: 10.1038/s41598-025-18186-5. PMID 41044147
- [Derived] Jensen IKB, Budtz-Jorgensen E, Lindh C, Roland CB, de Place Knudsen S, Bendix JM, Molsted S, Clausen TD, Stallknecht B, Mortensen OH, Lokkegaard E, Knudsen LE. Serum concentrations of per- and poly-fluoroalkyl substances (PFAS) in Danish pregnant women-temporal trends during pregnancy, correlations with partners, associations with physical activity, and blood lipid concentrations. Environ Health. 2025 Apr 2;24(1):16. doi: 10.1186/s12940-025-01170-x. PMID 40176054
- [Derived] Roland CB, Seyedhosseini P, Knudsen SP, Jessen AD, Jensen IKB, Bendix JM, van Hall G, Molsted S, Alomairah SA, Lokkegaard E, Stallknecht B, Clausen TD. Effects of prenatal exercise interventions on maternal body composition: A secondary analysis of the FitMum randomized controlled trial. PLoS One. 2024 Aug 1;19(8):e0308214. doi: 10.1371/journal.pone.0308214. eCollection 2024. PMID 39088510
- [Derived] Alomairah SA, Knudsen SP, Roland CB, Molsted S, Clausen TD, Bendix JM, Lokkegaard E, Jensen AK, Larsen JE, Jennum P, Stallknecht B. Effects of Two Physical Activity Interventions on Sleep and Sedentary Time in Pregnant Women. Int J Environ Res Public Health. 2023 Mar 31;20(7):5359. doi: 10.3390/ijerph20075359. PMID 37047973
- [Derived] Roland CB, Knudsen SD, Alomairah SA, Jessen AD, Jensen IKB, Braendstrup N, Molsted S, Jensen AK, Stallknecht B, Bendix JM, Clausen TD, Lokkegaard E. Effects of prenatal exercise on gestational weight gain, obstetric and neonatal outcomes: FitMum randomized controlled trial. BMC Pregnancy Childbirth. 2023 Mar 29;23(1):214. doi: 10.1186/s12884-023-05507-7. PMID 36991380
- [Derived] Knudsen SP, Alomairah SA, Roland CB, Jessen AD, Hergel IM, Clausen TD, Larsen JE, van Hall G, Jensen AK, Molsted S, Bendix JM, Lokkegaard E, Stallknecht B. Effects of Structured Supervised Exercise Training or Motivational Counseling on Pregnant Women's Physical Activity Level: FitMum - Randomized Controlled Trial. J Med Internet Res. 2022 Jul 20;24(7):e37699. doi: 10.2196/37699. PMID 35857356
- [Derived] Roland CB, Knudsen SP, Alomairah SA, Andersen AD, Bendix J, Clausen TD, Molsted S, Jensen AK, Teilmann G, Jespersen AP, Larsen JE, Hall GV, Andersen E, Barres R, Mortensen OH, Maindal HT, Tarnow L, Lokkegaard ECL, Stallknecht B. Structured supervised exercise training or motivational counselling during pregnancy on physical activity level and health of mother and offspring: FitMum study protocol. BMJ Open. 2021 Mar 19;11(3):e043671. doi: 10.1136/bmjopen-2020-043671. PMID 33741668

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03679130/SAP_000.pdf